CLINICAL TRIAL: NCT07375381
Title: Radiographic Assessment of the Correlation Between Maxillary Sinus Dimensions and Greater Palatine Canal Pathway in CBCT Images (A Retrospective Study).
Brief Title: CBCT Study of Maxillary Sinus Dimensions and Greater Palatine Canal Pathway: A Retrospective Analysis
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Lecturer, Faculty of Dentistry, Cairo University, Cairo University
Other Study IDs: 10/25
Record Dates: First submitted 2026-01-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Pneumatization
Keywords: pneumatization; CBCT; greater palatine canal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The CBCT-based radiographic evaluation will be used to identify, classify, and measure the anatomical parameters of the GPC and maxillary sinus. These data will serve as a pre-surgical diagnostic guide for clinicians when performing procedures involving the posterior maxilla.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years.
* Fully visible maxillary sinuses and complete GPC pathway in high-quality CBCT images.
* Scans free of motion or metallic artifacts.

Exclusion Criteria:

* History of maxillofacial trauma, orthognathic surgery, or pathology affecting the posterior maxilla.
* Craniofacial anomalies or syndromes.
* Poor-quality or incomplete scans.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult Egyptian patients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
To measure the height of the maxillary sinus in CBCT-reformatted panoramic views. | January 2026
  the height of the maxillary sinus will be measured in millimeters, in a coronal view.